CLINICAL TRIAL: NCT00459433
Title: The Right Intervention for the Right Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Back Research Center, Denmark (Other)
Collaborators: European Commission (Other)
Responsible Party: Bendt Johansen, MHS, The Back Research Center, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 258
Record Dates: First submitted 2007-04-10; First posted 2007-04-12 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Low Back Pain
Keywords: Low back pain; Return to work; Biopsychosocial; Screening; SMS; Non specific low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): psychosocial intervention
  Interventions: Procedure: Biopsychosocial intervention
- 2 (Active Comparator): Usual care
  Interventions: Procedure: Biopsychosocial intervention

INTERVENTIONS:
Procedure: Biopsychosocial intervention — Psychosocial versus usual care

SUMMARY:
Complicated and expensive interventions are used to treat unspecific low back pain and the intervention is not always targeted the patients specific problems.It is therefore not surprising that a large fraction of unspecific low back pain patients do not respond very well to the usual biopsychosocial intervention.

We would therefore like to identify the patients specific problems regarding the patients biomedical, psychological, and social needs.

DETAILED DESCRIPTION:
Two quality assurance investigations are performed in the The Back Research Center Clinic, where one is published in The Spine. The systematics of Health Technology Assessment was used to throw light on important indicators in relation to Health Technology aspects, patient aspects, organisational aspects and economical aspects. At 12 months follow up in 1999, approximately one third of the patients stated that their low back pain was unchanged or worse. In 2004 in a new investigation this fraction was larger. Therefore it seems relevant to be able to identify the patients early in their course in the back ambulatory.

A Norwegian project has shown that when one divides the patients into 3 levels of severity, then the interdisciplinary biopsychosocial intervention had best effect in the intermediary and severe groups. Conversely the mono disciplinary intervention had best effect on the least severe patient group.

Therefore we would like to combine elements from the typical clinical investigation with a screening for psychosocial factors in order to sort patients according to their individual needs.

Even though the bio-psycho-social elements are a coherent continuum one can arbitrarily combine them in 4 groups of increasing complexity.

* mainly biological
* both biological and psychological
* both biological and social
* both biological, psychological and social It is probably not good enough to give more or less the same type of somatic treatment to all unspecific low back pain patients. It is important to take into account all three elements, the severity of the elements, and the combination of elements. To be able to do this it is important to use a combination of screening instruments that can isolate and quantify the manifestations of the three elements in the patients.

ELIGIBILITY:
Inclusion Criteria:

* Unspecific low back pain
* Level of low back pain must be at least equal to leg pain
* Patients must have been sick listed during the past 12 months
* Age > 17 years and < than 60

Exclusion Criteria:

* Modic changes as seen on MRI
* Direct or progressive paresis or Cauda equina syndrome
* Known MB Bechterew or Sacroiliitis
* Suspicion of other serious malignancy
* Alcohol or medicine abuse
* A screening result of more than 30 in the Beck Depression Inventory

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Days on sick leave and days with low back pain problems measured every week by SMS questionnaire | 12 months

SECONDARY OUTCOMES:
Pain level | 12 months
Activity of daily living | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bendt Johansen, MHS, Principal Investigator — Affiliated with University of Southern Denmark
Locations (1):
- The Back Research Center, Ringe, Denmark

REFERENCES:
- [Background] Johansen B, Mainz J, Sabroe S, Manniche C, Leboeuf-Yde C. Quality improvement in an outpatient department for subacute low back pain patients: prospective surveillance by outcome and performance measures in a health technology assessment perspective. Spine (Phila Pa 1976). 2004 Apr 15;29(8):925-31. doi: 10.1097/00007632-200404150-00021. PMID 15082998
- [Background] Haldorsen EM, Grasdal AL, Skouen JS, Risa AE, Kronholm K, Ursin H. Is there a right treatment for a particular patient group? Comparison of ordinary treatment, light multidisciplinary treatment, and extensive multidisciplinary treatment for long-term sick-listed employees with musculoskeletal pain. Pain. 2002 Jan;95(1-2):49-63. doi: 10.1016/s0304-3959(01)00374-8. PMID 11790467